CLINICAL TRIAL: NCT02397720
Title: An Open-Label Phase II Study of Nivolumab (BMS-936558) in Combination With 5-Azacytidine (Vidaza) or Nivolumab With Ipilimumab in Combination With 5-Azacytidine for the Treatment of Patients With Refractory/ Relapsed Acute Myeloid Leukemia and Newly Diagnosed Older AML (> 65 Years) Patients
Brief Title: Nivolumab and Azacitidine With or Without Ipilimumab in Treating Patients With Refractory/Relapsed or Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0861; NCI-2015-00593 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0861 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Results first posted 2024-11-04 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Acute Bilineal Leukemia; Acute Biphenotypic Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; Ipilimumab; CTLA-4 Antigen; venetoclax; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1 A Lead-In (azacitidine, nivolumab) (Experimental): Patients receive azacitidine IV over 1 hour or SC on days 1-7 or days 1-4 and 7-9. Patients also receive nivolumab IV over 60 minutes on days 1 and 14 (courses 1-4) or on day 1 (course 5 and all subsequent courses). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Nivolumab
- Arm 2 A Lead-In (azacitidine, nivolumab, ipilimumab) (Experimental): Patients receive azacitidine and nivolumab as Arm I. Patients also receive ipilimumab IV over 90 minutes on day 1 and then every 6 or 12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Ipilimumab; Drug: Nivolumab
- Arm 1 B (azacitidine, nivolumab) (Experimental): Patients receive azacitidine IV over 1 hour or SC on days 1-7 or days 1-4 and 7-9. Patients also receive nivolumab IV over 60 minutes on days 1 and 14 (courses 1-4) or on day 1 (course 5 and all subsequent courses). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Nivolumab
- Arm 3 Lead-In (azacitidine, nivolumab, Venetoclax) (Experimental): Patients will receive therapy with nivolumab IV infusion on Day 8 and Day 22 (+/-3 days) of each 5-azacyidine cycle for first 4 cycles or until CR (whichever occurs earlier) followed by a maintenance regimen (one dose of nivolumab on Day 8 of each cycle of 5-azacytdine). Venetoclax will be administered orally daily on Days 1-21 of the first cycle; and Days 1-14 or Days 1-21 for subsequent cycles.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Nivolumab
- Arm 2 B (azacitidine, nivolumab, ipilimumab) (Experimental): Patients receive azacitidine and nivolumab as Arm I. Patients also receive ipilimumab IV over 90 minutes on day 1 and then every 6 or 12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Ipilimumab; Drug: Nivolumab
- Arm 3 (azacitidine, nivolumab, Venetoclax) (Experimental): Patients will receive therapy with nivolumab IV infusion on Day 8 and Day 22 (+/-3 days) of each 5-azacyidine cycle for first 4 cycles or until CR (whichever occurs earlier) followed by a maintenance regimen (one dose of nivolumab on Day 8 of each cycle of 5-azacytdine). Venetoclax will be administered orally daily on Days 1-21 of the first cycle; and Days 1-14 or Days 1-21 for subsequent cycles.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Nivolumab

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Ipilimumab
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm 2 A Lead-In (azacitidine, nivolumab, ipilimumab); Arm 2 B (azacitidine, nivolumab, ipilimumab)
Drug: Venetoclax — Given Orally
  Other Names: ABT-199; GDC-0199
  Arms: Arm 3 (azacitidine, nivolumab, Venetoclax); Arm 3 Lead-In (azacitidine, nivolumab, Venetoclax)
Drug: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This will be a phase II, open-label, non-randomized study with a safety lead-in phase. There are 3 Arms in this study each with 2 parts. If you are eligible, you will be assigned to an Arm and a part when you join the study. In each arm, you will receive a different combination of study drugs: Arm 1: nivolumab and azacitidine, Ih Arm 2: nivolumab, azacitidine, and ipilimumab, Arm 3: nivolumab, azacitidine, and venetoclax.

There are 2 parts in each arm: Part A (dose escalation) and Part B (dose expansion).

The goal of Part A of this clinical research study is to find the highest tolerable dose of the study drugs (nivolumab, azacitidine, ipilimumab, and/or venetoclax) that can be given to patients with AML. The goal of Part B of this study is to learn if the dose found in Part A can help to control AML.

DETAILED DESCRIPTION:
Arm 1 Up to 5 groups of up to 6 participants will be enrolled in Part A of the study, and up to 110 participants will be enrolled in Part B of the study. If you are enrolled in Part A of the study, the dose of nivolumab and azacitidine you receive will depend on when you joined this study. The first group of participants will receive the starting dose levels of nivolumab and azacitidine. If intolerable side effects are seen, the next group may receive a lower dose level of nivolumab and/or azacitidine. This will continue until the highest tolerable combination dose is found.

If you are enrolled in Part B, you will receive nivolumab and azacitidine at the highest dose that was tolerated in Part A.

Arm 2 Up to 4 groups of up to 6 participants will be enrolled in Part A of the study, and up to 84 participants will be enrolled in Part B of the study. If you are enrolled in Part A of the study, the dose of nivolumab, azacitidine, and ipilimumab you receive will depend on when you joined this study. The first group of participants will receive the starting dose levels of nivolumab, azacitidine and ipilimumab. If intolerable side effects are seen, the next group may receive a lower dose level of nivolumab, azacitidine and/or ipilimumab. This will continue until the highest tolerable combination dose is found. If you are enrolled in Part B, you will receive nivolumab, azacitidine, and ipilimumab at the highest dose that was tolerated in Part A.

Arm 3 About 6-18 participants will be enrolled in Part A and up to 60 participants will be enrolled in Part B. If you are enrolled in Part A of the study, the dose of nivolumab, azacitidine, and venetoclax you receive will depend on when you joined this study. The first group of participants will receive the starting dose levels of nivolumab, azacitidine and venetoclax. If intolerable side effects are seen, the next group may receive a lower dose level of nivolumab, azacitidine and/or venetoclax. This will continue until the highest tolerable combination dose is found. If you are enrolled in Part B, you will receive nivolumab, azacitidine, and venetoclax at the highest dose that was tolerated in Part A.

ELIGIBILITY:
Inclusion Criteria:

* ARM 1 SALVAGE COHORT: Patients with AML or biphenotypic or bilineage leukemia who have failed prior therapy; patients with AML should have failed prior therapy or have relapsed after prior therapy will be eligible for Arm 1;
* ARM 2 SALVAGE COHORT: Patients with AML who have failed up to one prior salvage therapy (i.e. salvage 1 or 2 status) will be eligible for Arm 2 relapse cohort; allogeneic stem cell transplant for patients in remission at the time of stem cell transplant will not be considered a salvage regimen; similarly, hydroxyurea if used alone will not be considered a salvage regimen
* ARM 1 AND 2 FRONT LINE OLDER COHORT: Patients age 65 years and above with previously untreated AML who are unfit for or decline standard induction therapy; prior therapy with hydroxyurea, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors), or hematopoietic growth factors is allowed, however prior therapy with chemotherapy agents for the disease under study is not allowed; patients may have received one dose of cytarabine (up to 2 g/m2 administered at presentation for control) of hyperleucocytosis
* Patients with myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) who received therapy for the MDS or CMML and progress to AML are eligible at the time of diagnosis of AML regardless any prior therapy for MDS or CMML; the World Health Organization (WHO) classification will be used for AML; prior therapy for MDS or CMML will not be considered as a prior therapy for AML, hence such patients will be considered as frontline AML and eligible for the frontline elderly cohort
* Prior therapy with hydroxyurea, chemotherapy, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors), or hematopoietic growth factors is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 2 times upper limit of normal (x ULN) (=< 3 x ULN if considered to be due to leukemic involvement or Gilbert's syndrome)
* Aspartate aminotransferase or alanine aminotransferase =< 2.5 x ULN (=< 5.0 x ULN if considered to be due to leukemic involvement)
* Serum creatinine =< 2 x ULN or glomerular filtration rate (GFR) >= 50
* Patients must provide written informed consent
* In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of 5-azacytidine and nivolumab will be at least 2 weeks OR at least 5 half-lives for cytotoxic/noncytotoxic agents; the half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochure's, or drug-administration manuals) and will be documented in the protocol eligibility document; since the effect of both nivolumab and 5-azacytidine may be delayed; use of one dose of cytarabine (up to 2 g/m2) or hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and during the study treatment; concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment; males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment; adequate methods of contraception include: total abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception; female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment; male sterilization (at least 6 months prior to screening); for female patients on the study, the vasectomized male partner should be the sole partner for that patient
* Combination of any of the two following

  * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository; in case of use of oral contraception, women should have been stable on the same pill before taking study treatment; note: oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Patients with graft versus host disease (GVHD) active < grade 2 who are on a stable dose of immunosuppressive therapy (tacrolimus, cyclosporine, or other) for > 2 weeks will be included; Note: subjects may be using systemic corticosteroids or topical or inhaled corticosteroids

Exclusion Criteria:

* Patients with known allergy or hypersensitivity to nivolumab, ipilimumab, 5-azacytidine, or any of their components
* Patients with a known history of severe interstitial lung disease or severe pneumonitis or active pneumonitis that is uncontrolled in the opinion of the treating physician
* Patients who have previously been treated with nivolumab and/or ipilimumab in combination with 5-azacytidine will be excluded
* Patients with a known history of any of the following autoimmune diseases are excluded:

  * Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis)
  * Patients with a history of rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis (e.g., Wegener's granulomatosis)
* Patients with organ allografts (such as renal transplant) are excluded
* Patients with active GVHD > grade 2 will be excluded; patients with recent increase in the immunosuppressive medication dose within last 2 weeks to control GVHD will not be included; patients with grade 1 or lower GVHD on =< 10 mg prednisone without any additional immunosuppressive therapies (tacrolimus, prograf, etc) will be eligible
* Patients with symptomatic CNS leukemia or patients with poorly controlled CNS leukemia
* Active and uncontrolled disease/(active uncontrolled infection, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association [NYHA] class III/IV, clinically significant and uncontrolled arrhythmia) as judged by the treating physician
* Patients with known human immunodeficiency virus seropositivity will be excluded
* Known to be positive for hepatitis B by surface antigen expression; known to have active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months)
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator
* Patients unwilling or unable to comply with the protocol
* Pregnant or breastfeeding
* Acute promyelocytic leukemia (APL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Root JL, Desai PN, Ly C, Wang B, Jelloul FZ, Zhou J, Mackay S, Alfayez M, Matthews J, Pierce S, Reville PK, Daver N, Abbas HA. Single-Cell CD4 and CD8 T-Cell Secretome Profiling Reveals Temporal and Niche Differences in Acute Myeloid Leukemia Following Immune Checkpoint Blockade Therapy. Cancer Res Commun. 2024 Mar 6;4(3):671-681. doi: 10.1158/2767-9764.CRC-23-0402. PMID 38391202
- [Derived] El Hussein S, Daver N, Liu JL, Kornblau S, Fang H, Konoplev S, Kantarjian H, Khoury JD. Microsatellite Instability Assessment by Immunohistochemistry in Acute Myeloid Leukemia: A Reappraisal and Review of the Literature. Clin Lymphoma Myeloma Leuk. 2022 Jun;22(6):e386-e391. doi: 10.1016/j.clml.2021.12.004. Epub 2021 Dec 9. PMID 34980577
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab); Arm 2 B (Azacitidine, Nivolumab, Ipilimumab): Patients receive azacitidine and nivolumab as Arm I. Patients also receive ipilimumab IV over 90 minutes on day 1 and then every 6 or 12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Azacitidine: Given SC or IV
  Ipilimumab
  Nivolumab: Given IV
- Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax); Arm 3 B (Azacitidine, Nivolumab, Venetoclax): Patients will receive therapy with nivolumab IV infusion on Day 8 and Day 22 (+/-3 days) of each 5-azacyidine cycle for first 4 cycles or until CR (whichever occurs earlier) followed by a maintenance regimen (one dose of nivolumab on Day 8 of each cycle of 5-azacytdine). Venetoclax will be administered orally daily on Days 1-21 of the first cycle; and Days 1-14 or Days 1-21 for subsequent cycles.
  Azacitidine: Given SC or IV
  Venetoclax: Given Orally
  Nivolumab: Given IV
Period: Overall Study
Arm/Group | Arm 1 A Lead-In (Azacitidine, Nivolumab) | Arm 1 B (Azacitidine, Nivolumab) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) | Arm 2 B (Azacitidine, Nivolumab, Ipilimumab) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax) | Arm 3 B (Azacitidine, Nivolumab, Venetoclax)
Started | 6 | 85 | 6 | 47 | 6 | 0 (There were Zero participants enrolled on Arm 3 B due to no responses in the lead in phase.)
Completed | 6 | 85 | 6 | 47 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were Zero participants enrolled on Arm 3 B due to no responses in the lead in phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 A Lead-In (Azacitidine, Nivolumab) | Arm 1 B (Azacitidine, Nivolumab) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) | Arm 2 B (Azacitidine, Nivolumab, Ipilimumab) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax) | Arm 3 B (Azacitidine, Nivolumab, Venetoclax) | Total
Number analyzed (Participants) | 6 | 85 | 6 | 47 | 6 | 0 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 25 | 3 | 21 | 2 | 0 | 54
  >=65 years | 3 | 60 | 3 | 26 | 4 | 0 | 96
Age, Continuous [Median (Full Range); unit: years] | 60 [45 to 73] | 71 [22 to 90] | 66 [25 to 77] | 66 [21 to 83] | 67 [48 to 72] |  | 69 [21 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 25 | 3 | 18 | 3 |  | 50
  Male | 5 | 60 | 3 | 29 | 3 |  | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 |  | 0
  Asian | 0 | 1 | 0 | 1 | 0 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 1 | 5 | 1 | 1 | 0 |  | 8
  White | 4 | 70 | 5 | 43 | 5 |  | 127
  More than one race | 0 | 0 | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 1 | 9 | 0 | 2 | 1 |  | 13
Region of Enrollment [Number; unit: participants]
  United States | 6 | 85 | 6 | 47 | 6 |  | 150

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of 5-azacytidine in the Combination of Nivolumab With Dihydro-5-azacytidine
Description: The maximum tolerated dose is defined as the highest dose level of 5-azacitidine with < 2 out of 6 patients experiencing a dose limiting toxicity during the first 28 days of treatment. The starting dose level for Azacitidine is 75 mg/m^2 and the starting dose level for Nivolumab is 3.0 mg/kg.
Time Frame: Up to 28 days
Population: All participants were treated at dose level 0, the starting dose.
Measure: Number; unit: Mg/m^2
Arm/Group | Arm 1 A Lead-In (Azacitidine, Nivolumab) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax)
Number analyzed (Participants) | 6 | 6 | 6
Mg/m^2 | 75 | 75 | 75

2. Primary Outcome: Participants With a Response
Description: Responders are patients who obtain a Complete Remission (CR), Complete Remission with Incomplete blood count recovery CRi, Complete Remission with Incomplete Platelet Recovery (CRp) or Partial Remission (PR), with or without cytogenetic response, hematologic improvements (HI), and morphologic leukemia-free state. CR is counts of 0 circulating blasts, Neutrophil count of >/= 1.0 x 10^9/L, Platelet count >/= 100 x 10 ^9/L. Bone marrow </= 5% blasts, No auer rods, No extramedullary disease. CRp is patients who have achieved a CR except for incomplete platelet recovery (<100 x 10^9/L). CRi is counts of 0 circulating blasts, Neutrophil count of >/= 1.0 x 10^9/L OR Platelet count >/= 100 x 10 ^9/L. PR is All CR criteria if abnormal before treatment except >/= 50% reduction in bone marrow blast but still >5%. morphologic leukemia-free state is Bone marrow: </=5% myeloblasts. HI is Hematologic response must be described by the number of positively affected cell lines.
Time Frame: Up to 7 years, 6 months
Population: There were Zero participants enrolled on Arm 3 B due to no responses in the lead in phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 A Lead-In (Azacitidine, Nivolumab) | Arm 1 B (Azacitidine, Nivolumab) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) | Arm 2 B (Azacitidine, Nivolumab, Ipilimumab) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax)
Number analyzed (Participants) | 6 | 85 | 6 | 47 | 6
Participants | 2 | 34 | 2 | 13 | 4

3. Secondary Outcome: Disease-free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 7 years, 6 months
Population: There were Zero participants enrolled on Arm 3 B due to no responses in the lead in phase.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 1 A Lead-In (Azacitidine, Nivolumab) | Arm 1 B (Azacitidine, Nivolumab) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) | Arm 2 B (Azacitidine, Nivolumab, Ipilimumab) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax)
Number analyzed (Participants) | 2 | 34 | 2 | 13 | 2
Months | 3.0 [2.9 to 3.1] | 7.1 [0.4 to 90.0] | 4.1 [0.1 to 8.2] | 2.0 [0.0 to 5.7] | 2.9 [0.9 to 4.9]

4. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 7 years, 6 months
Population: There were Zero participants enrolled on Arm 3 B due to no responses in the lead in phase.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 1 A Lead-In (Azacitidine, Nivolumab) | Arm 1 B (Azacitidine, Nivolumab) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) | Arm 2 B (Azacitidine, Nivolumab, Ipilimumab) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax)
Number analyzed (Participants) | 6 | 85 | 6 | 47 | 6
Months | 5.9 [3.5 to 16.2] | 6.6 [0.3 to 90.0] | 8.3 [3.1 to 32.4] | 6.7 [0.4 to 71.5] | 1.4 [1.0 to 8.8]

5. Secondary Outcome: Progression-free Survival
Description: Time from date of treatment start until the date of progression or death from leukemia.
Time Frame: Up to 7 years, 6 months
Population: There were Zero participants enrolled on Arm 3 B due to no responses in the lead in phase.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 1 A Lead-In (Azacitidine, Nivolumab) | Arm 1 B (Azacitidine, Nivolumab) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) | Arm 2 B (Azacitidine, Nivolumab, Ipilimumab) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax)
Number analyzed (Participants) | 6 | 85 | 6 | 47 | 6
Months | 3.5 [2.3 to 16.2] | 3.5 [0.3 to 90.0] | 3.2 [1.6 to 11.9] | 3.6 [0.2 to 15.8] | 1.3 [1.0 to 8.8]

6. Primary Outcome: Maximum Tolerated Dose of Nivolumab in the Combination of Nivolumab With Dihydro-5-azacytidine
Description: The maximum tolerated dose is defined as the highest dose level of nivolumab with < 2 out of 6 patients experiencing a dose limiting toxicity during the first 28 days of treatment. The starting dose level for Azacitidine is 75 mg/m^2 and the starting dose level for Nivolumab is 3.0 mg/kg.
Time Frame: Up to 28 days
Population: All participants were treated at dose level 0, the starting dose.
Measure: Number; unit: mg/kg
Arm/Group | Arm 1 A Lead-In (Azacitidine, Nivolumab) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax)
Number analyzed (Participants) | 6 | 6 | 6
mg/kg | 3 | 3 | 3

ADVERSE EVENTS:
Time Frame: Up to 7 years, 6 months
Description: There were Zero participants enrolled on Arm 3 B due to no responses in the lead in phase.
Arm/Group | Arm 1 A Lead-In (Azacitidine, Nivolumab) | Arm 1 B (Azacitidine, Nivolumab) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) | Arm 2 B (Azacitidine, Nivolumab, Ipilimumab) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax) | Arm 3 B (Azacitidine, Nivolumab, Venetoclax)
All-Cause Mortality (participants affected / at risk) | 1/6 | 16/85 | 1/6 | 5/47 | 1/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 6/6 | 57/85 | 2/6 | 33/47 | 5/6 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 62/85 | 5/6 | 25/47 | 4/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 A Lead-In (Azacitidine, Nivolumab) (N=6) | Arm 1 B (Azacitidine, Nivolumab) (N=85) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) (N=6) | Arm 2 B (Azacitidine, Nivolumab, Ipilimumab) (N=47) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax) (N=6) | Arm 3 B (Azacitidine, Nivolumab, Venetoclax) (N=0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 25 (36) | 2 (5) | 15 (22) | 3 (3) | 0 (0)
General disorders and administration site conditions (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (4) | 32 (45) | 1 (1) | 15 (25) | 2 (3) | 0 (0)
Lumbar Spine Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 10 (10) | 1 (1) | 6 (6) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Investigations (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi organ failure (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 8 (11) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures Biliary Drain Removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 A Lead-In (Azacitidine, Nivolumab) (N=6) | Arm 1 B (Azacitidine, Nivolumab) (N=85) | Arm 2 A Lead-In (Azacitidine, Nivolumab, Ipilimumab) (N=6) | Arm 2 B (Azacitidine, Nivolumab, Ipilimumab) (N=47) | Arm 3 A Lead-In (Azacitidine, Nivolumab, Venetoclax) (N=6) | Arm 3 B (Azacitidine, Nivolumab, Venetoclax) (N=0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (4) | 0 (0) | 5 (7) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Benign Prostatic Hyperplasia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelosuppression (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 17 (22) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 18 (28) | 0 (0) | 2 (5) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Edema (General disorders) | 3 (6) | 6 (7) | 0 (0) | 4 (6) | 1 (1) | 0 (0)
Endocrine disorders (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Disorders (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 13 (21) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 3 (4) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (5) | 3 (3) | 0 (0)
General disorders and administration site conditions (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (General disorders) | 2 (3) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 5 (8) | 2 (2) | 7 (13) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (7) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6) | 0 (0) | 3 (5) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 6 (7) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (6) | 10 (12) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Investigations (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 8 (9) | 1 (4) | 5 (6) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 10 (17) | 0 (0) | 2 (4) | 3 (3) | 0 (0)
Nervous system disorders (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 7 (10) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (10) | 10 (32) | 1 (1) | 6 (10) | 3 (8) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pneumonitis (Infections and infestations) | 0 (0) | 6 (8) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (9) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (5) | 2 (2) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 7 (8) | 0 (0) | 3 (5) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 (7) | 6 (10) | 0 (0) | 5 (10) | 2 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (10) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT02397720/Prot_SAP_000.pdf